CLINICAL TRIAL: NCT05033873
Title: Comparison of Universal Exercise Unit Therapy With Sling Exercise Therapy on Lower Limb Kinematics in Chronic Stroke Patients
Brief Title: Universal Exercise Unit Therapy With Sling Exercise Therapy on Lower Limb Kinematics in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/1108
Record Dates: First submitted 2021-06-26; First posted 2021-09-05 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Chronic Stroke
Keywords: Motion analysis; Universal exercise unit; Sling exercise therapy; Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Universal Exercise Unit Therapy (UEU) (Experimental): This experimental group will be given universal exercise unit therapy.
  Interventions: Other: Universal Exercise Unit Therapy (UEU)
- Group B: Sling Exercise Therapy (SET) (Experimental): This experimental group will be given sling exercise therapy
  Interventions: Other: Sling Exercise Therapt (SET)
- Group C: Control Group (Other): Control group will be given routine physical therapy
  Interventions: Other: Routine Physical Therapy / Control Group

INTERVENTIONS:
Other: Universal Exercise Unit Therapy (UEU) — Standing, walk standing, half standing, kneel standing, half kneel standing, quadruped position, three point quadruped , alternative quadruped , transitions, walking all these will be done in Universal Exercise Unit with a standardized protocol regimen.
  Other Names: Group A
  Arms: Group A: Universal Exercise Unit Therapy (UEU)
Other: Sling Exercise Therapt (SET) — 1. The patient's bilateral knee joints/feet will be suspended by a rope belt, and then the patient's pelvis will be elevated and maintained in supine or lateral position, adding flexion and extension training to lower limb if permitted.
  2. In supine or lateral position, with patient's head, trunk and pelvis fixed, the therapist will use appropriate elastic bands to assist patient's limbs to do passive-power assisted-power resistance training in all directions (bending, stretch, outreach, and adduction).
  3. The patient's chest and abdomen will be suspended by a wide elastic band, positioned him-self in the prone position with the fulcrum of bilateral elbows and knees, and then the torso swayed in all directions, therapists could assist
  4. Target elbow and wrist will be suspended, according to the patient's ability to do passive/active open and close chain movement
  Other Names: Group B
  Arms: Group B: Sling Exercise Therapy (SET)
Other: Routine Physical Therapy / Control Group — Control group will receive routine physiotherapy with duration one hour including
  * Active and passive joint movement
  * Muscle strength training
  * Bridging exercises
  * Balance training in sitting and standing positions, according to the patients' functional state.
  * Weight bearing exercises on affected Limbs
  Other Names: Group C
  Arms: Group C: Control Group

SUMMARY:
Stroke occurred when blood supply to brain or a part of brain is disturbed due to clot (ischaemic stroke) or due rupture of small vessels (hemorrhagic stroke) in brain and causes bleeding in brain cells. The prevalence of stroke was 1.2 % (1200/100,000) in Pakistan, 3.1% in China and it is 44.29 to 559/100,000 in different parts of the world. Leading cause of stroke is hypertension. The aim of study will be to compare universal exercise unit therapy with sling exercise therapy on lower limb kinematics, disability, balance and quality of life in chronic stroke patients.

DETAILED DESCRIPTION:
This will be randomized controlled trial. Study will be conducted at Khawaja Arshed Hospital Sargodha. Duration of intervention will be 08 weeks, 5 sessions in a week, total 40 sessions. Duration of single session will be one hour. A convenient sample of n patients fulfilling the inclusion and exclusion criteria will be selected from in-patient settings of various hospitals from the city Sargodha and will be allocated randomly into three groups equally after taking informed consent. Group A will obtain Universal Exercise Unit Therapy. Group B will obtain Sling Exercise Therapy and Group C will be control and will receive routine physical therapy. Outcome will be measured at baseline, 04 weeks and 08 weeks. Outcome measurement tools will be Berg balance scale, Barthel index, Short form 12 (SF-12), Trunk impairment scale, functional reach test and smart phone motion analysis for lower limb kinematics. Scores will be measure in mean and SD. Results of intervention will be comparing by using one way ANOVA by using IBM SPSS version 21.0

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic (course of disease at least six month)
* Recently discharge from in-patients setting with in 06 month of onset
* Hemiplegia (either right or left)
* Both gender
* Age between 30 to 70
* Medically stable
* No balance disorders before this stroke.
* History of mental
* illness or severe cognitive impairment (MINI-MENTAL SCALE SCORE > 25)

Exclusion Criteria:

* Stroke Patient with complication like shoulder hand syndrome, adhesive capsulitis or shoulder partial dislocation
* Stroke patients with behavioral issue, significant cognitive deficit
* Patients with arthritis and fracture
* Chronic stroke with deformities
* Serious viscera dysfunction, such as cardiovascular system,
* Lung, liver and kidney
* History of mental
* Illness or severe cognitive impairment (MINI-MENTAL SCALE SCORE > 25)
* Audio-visual understanding
* obstacle, unable to cooperate with instructions;
* Infection and ulcer skin

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
THE BERG BALANCE SCALE: (BALANCE FUNCTION) | 2 months
  This scale will be used to check the balance of the patients during the functional activities. Scale consists of 14 tasks and each task can be scored between 0 and 4. Overall balance score ranges from 0 to 56. 0 score is showing severely damage balance and 56 score is showing excellent balance. A score below 40 indicate the risk of falling in particular function.
BARTHEL INDEX: (FUNCTIONAL ABILITY) | 2 months
  This index is used to measure the activities of daily life, having total 10 items and can be scored from 0 to 100.
SHORT FORM 12 (SF-12): (QUALITY OF LIFE) | 2 months
  This survey contains 12 items divided into eight domains: physical function (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social function (SF), role-emotional (RE), and mental health (MH). According to the calculation formula, raw scores were converted into final scores. As scores increased, health status and quality of life increased for the subject.
SMART PHONE MOTION ANALYSIS FOR LOWER LIMB KINEMATICS DURING WALKING | 2 months
  Sagittal plane hip, knee, and ankle angle and rear foot eversion will be assessed by using the Coach's Eye Smart phone application
FUNCTIONAL REACH TEST | 2months
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task. In standing, measures the distance between the lengths of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.
TRUNK IMPAIRMENT SCALE | 2 Months
  The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Study Chair — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajkumar S, Chandra SB. Recent advances in treatment of cerebral ischemic stroke. Medicine. 2021;10(1):1.
- [Background] Busl KM, Greer DM. Hypoxic-ischemic brain injury: pathophysiology, neuropathology and mechanisms. NeuroRehabilitation. 2010;26(1):5-13. doi: 10.3233/NRE-2010-0531. PMID 20130351
- [Background] Sherin A, Ul-Haq Z, Fazid S, Shah BH, Khattak MI, Nabi F. Prevalence of stroke in Pakistan: Findings from Khyber Pakhtunkhwa integrated population health survey (KP-IPHS) 2016-17. Pak J Med Sci. 2020 Nov-Dec;36(7):1435-1440. doi: 10.12669/pjms.36.7.2824. PMID 33235553
- [Background] Yi X, Luo H, Zhou J, Yu M, Chen X, Tan L, Wei W, Li J. Prevalence of stroke and stroke related risk factors: a population based cross sectional survey in southwestern China. BMC Neurol. 2020 Jan 7;20(1):5. doi: 10.1186/s12883-019-1592-z. PMID 31910820
- [Background] Kamalakannan S, Gudlavalleti ASV, Gudlavalleti VSM, Goenka S, Kuper H. Incidence & prevalence of stroke in India: A systematic review. Indian J Med Res. 2017 Aug;146(2):175-185. doi: 10.4103/ijmr.IJMR_516_15. PMID 29265018
- [Background] Venketasubramanian N, Yoon BW, Pandian J, Navarro JC. Stroke Epidemiology in South, East, and South-East Asia: A Review. J Stroke. 2017 Sep;19(3):286-294. doi: 10.5853/jos.2017.00234. Epub 2017 Sep 29. PMID 29037005
- [Background] Hussein ZA. Strength training versus chest physical therapy on pulmonary functions in children with Down syndrome. Egyptian Journal of Medical Human Genetics. 2017;18(1):35-9.
- [Background] Wooten A. Universal Exercise Unit for Treatment of a Child Following Hemispherectomy: A Case Report. 2017.
- [Background] Salim ASM. Effect of universal exercise unit on standing in spastic diaplegia. 2013.
- [Background] Olama KA, Elnahhas AM, Rajab SH. Effect of universal exercise unit on balance in children with spastic Diplegia.